CLINICAL TRIAL: NCT00282828
Title: Improving Outcomes in Pharmacotherapy of Social Phobia
Brief Title: Improving Treatment Outcomes in Pharmacotherapy of Generalized Social Anxiety Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Mark H. Pollack, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01MH070919 (NIH); R01MH070919 (NIH); PA-01-123; DSIR 83-ATAS
Record Dates: First submitted 2006-01-25; First posted 2006-01-27 (Estimated); Results first posted 2013-10-14 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-08

CONDITIONS: Social Phobia
Keywords: Social Anxiety Disorder; Pharmacotherapy; Genetics; Treatment Refractory
MeSH Terms: conditions — Phobia, Social | interventions — Sertraline; Venlafaxine Hydrochloride; Clonazepam

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sertraline & Clonazepam (Experimental): Phase I non-responders randomized to this group remained on sertraline at the same dose level as at entry into Phase 2 with the addition of clonazepam up to 3.0mg per day.
  Dosing was flexible, permitting clinicians to slow or suspend the titration of the medication because of side effects or response, but patients had to receive no less than 0.5mg of clonazepam per day in order to remain in the study.
  Interventions: Drug: Sertraline; Drug: Clonazepam
- Venlafaxine (Experimental): Phase I non-responders randomized to this group switched to venlafaxine with flexible titration up to 225 mg per day.
  Dosing was flexible, permitting clinicians to slow or suspend the titration of the medication because of side effects or response, but patients had to receive no less than 75 mg venlafaxine per day in order to remain in the study.
  Interventions: Drug: Venlafaxine
- Sertraline & Placebo (Experimental): Phase I non-responders randomized to this group remained on sertraline at the same dose level as at entry into Phase 2 with the addition of placebo.
  Dosing was flexible, permitting clinicians to slow or suspend the titration of the medication because of side effects or response, but patients had to receive no less than 1 capsule of placebo per day in order to remain in the study.
  Interventions: Drug: Sertraline; Drug: Placebo

INTERVENTIONS:
Drug: Sertraline
  Arms: Sertraline & Clonazepam; Sertraline & Placebo
Drug: Venlafaxine
  Arms: Venlafaxine
Drug: Placebo
  Arms: Sertraline & Placebo
Drug: Clonazepam
  Arms: Sertraline & Clonazepam

SUMMARY:
This study will compare the effectiveness of either adding clonazepam or placebo to standard treatment or switching to venlafaxine in treating generalized social anxiety disorder in individuals who have not responded to treatment with sertraline.

DETAILED DESCRIPTION:
Generalized social anxiety disorder (GSAD) is one of the most common psychiatric disorders, and often causes significant distress and dysfunction in affected individuals. Although currently available treatments for GSAD are effective, most individuals have residual symptoms after initial psychosocial or psychopharmacologic intervention. Further treatment is necessary for such individuals, but sufficient research has not been done to guide clinicians on what the safest and most effective next step may be. This study will compare the effectiveness of either combining clonazepam or placebo with sertraline or completely switching to venlafaxine in treating GSAD in individuals who have not responded to treatment with sertraline. This study will also examine predictors of treatment response, including factors such as age at disease onset, duration of illness, comorbidities, and genes that influence serotonin and catecholamine metabolism.

Participants in this double-blind study will first partake in an initial 10-week phase in which they will be treated with sertraline. Participants who do not respond to sertraline treatment will proceed to phase two of the study, in which they will be randomly assigned to one of three treatment groups. One group will receive both sertraline and clonazepam, another group will receive both sertraline and placebo, and the third group will receive only venlafaxine. All treatments will continue for 12 weeks. Sertraline and venlafaxine are both FDA-approved for the treatment of GSAD. Clonazepam is widely used for the treatment of anxiety, but is not FDA-approved for the treatment of GSAD. All participants will attend weekly study visits at Weeks 1, 2, 4, 6, 8, and 10. Participants who continue into phase two will attend weekly study visits at Weeks 11-14, 16, 18, 20, and 22. Symptom remission rates and post-treatment social phobia severity will be assessed at Week 22.

ELIGIBILITY:
Inclusion Criteria:

* Primary psychiatric diagnosis of GSAD as defined by DSM-IV criteria and a score above 60 on the LSAS
* Agrees to use an effective form of contraception throughout the study

Exclusion Criteria:

* Clinically significant abnormalities found upon physical examination, electrocardiogram, and laboratory tests
* History of more than two unsuccessful, adequate treatment trials, indicated by a lack of response to over 10 weeks of any of the following: SSRIs (e.g., 40 mg of paroxetine or its equivalent per day); benzodiazepine (e.g. at least 2.5 mg of clonazepam per day) plus antidepressant (adequate dose as above); monoamine oxidase inhibitors (e.g., 60 mg of phenelzine or its equivalent per day); or a single failed trial of over 10 weeks of venlafaxine ( at least 150 mg per day)
* Pregnant or breastfeeding
* Simultaneous use of other psychotropic medications, with the exception of psychostimulants to treat ADHD; participants must discontinue regular benzodiazepine or antidepressant therapy at least two weeks (5 weeks for fluoxetine) prior to study entry; beta-blockers must be discontinued unless they are indicated medically (e.g., for hypertension)
* DSM-IV diagnosis of any of the following: lifetime history of schizophrenia or any other psychosis, mental retardation, organic medical disorder, bipolar disorder, or obsessive compulsive disorder; eating disorder in the past 6 months; alcohol or substance abuse in the past 3 months or dependence within the past 6 months (entry of participants with major depression, dysthymia, panic disorder, generalized anxiety disorder, or post-traumatic stress disorder will be permitted if the social anxiety disorder is judged to be the predominant disorder)
* Significant suicidal ideation as indicated by a score greater than 3 on the Montgomery-Asberg Depression Rating Scale or suicidal behaviors within 6 months prior to study entry
* Significant personality dysfunction that could interfere with study participation
* Serious medical illness or instability for which hospitalization may be likely during the study
* Seizure disorders, with the exception of a childhood history of isolated, non-recurrent febrile seizures
* Any concurrent psychotherapy initiated within 3 months of study entry, or ongoing psychotherapy of any duration directed specifically toward treatment of GSAD (prohibited psychotherapy includes cognitive behavioral therapy or psychodynamic therapy that focuses on exploring specific, dynamic causes of the phobic symptomatology and that provides management skills; general supportive therapy for more than 3 months is acceptable)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2006-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark H. Pollack, MD, Principal Investigator — Massachusetts General Hospital; Murray B. Stein, MD, MPH, Principal Investigator — University of California San Deigo; Michael Van Ameringen, MD, FRCPC, Principal Investigator — Anxiety Disorders Clinic McMaster University Medical Centre
Locations (3):
- United States (2):
  - University of California San Diego, La Jolla, California
  - Center for Anxiety and Traumatic Stress Disorders, Boston, Massachusetts
- McMaster University Medical Centre Anxiety Disorders Clinic, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Pollack MH, Van Ameringen M, Simon NM, Worthington JW, Hoge EA, Keshaviah A, Stein MB. A double-blind randomized controlled trial of augmentation and switch strategies for refractory social anxiety disorder. Am J Psychiatry. 2014 Jan;171(1):44-53. doi: 10.1176/appi.ajp.2013.12101353. PMID 24399428
- See also: Click here for the Anxiety Disorders Association of America website — http://www.adaa.org
- See also: Please click here for UCSD Anxiety and Traumatic Stress Disorders Research Program — http://www.veryshy.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this study began in 2006 at the Massachusetts General Hospital, the University of California San Diego, and the Anxiety Disorders Clinic, McMaster University Medical Centre. Through approved recruitment methods, 397 patients with Generalized Social Anxiety Disorder (GSAD) were enrolled in Phase I of the study (open sertraline).
Pre-assignment Details: Among the 397 patients enrolled in Phase I of the study, 295 patients entered Phase II. A total of 181 (61%) of the patients who began Phase II were non-responders at week 10 (LSAS>50), and were therefore randomized to receive 12 weeks of treatment in one of three treatment arms (sertraline plus clonazepam, venlafaxine, or sertraline plus placebo).
Groups:
- Sertraline and Clonazepam: Phase I non-responders randomized to this group remained on sertraline with the addition of clonazepam up to 3.0mg/d.
- Venlafaxine: Phase I non-responders randomized to this group switched to venlafaxine with flexible titration up to 225 mg/d.
- Sertraline and Placebo: Phase I non-responders randomized to this group received prolonged sertraline and placebo.
Period: Overall Study
Arm/Group | Sertraline and Clonazepam | Venlafaxine | Sertraline and Placebo
Started | 63 | 59 | 59
Completed | 57 | 47 | 50
Not Completed | 6 | 12 | 9

BASELINE CHARACTERISTICS:
Groups:
- Sertraline and Clonazepam: Participants will take both sertraline and clonazepam
- Venlafaxine: Participants will take venlafaxine only
- Sertraline and Placebo: Participants will take both sertraline and placebo
- Total: Total of all reporting groups
Arm/Group | Sertraline and Clonazepam | Venlafaxine | Sertraline and Placebo | Total
Number analyzed (Participants) | 63 | 59 | 59 | 181
Age Continuous [Mean (Standard Deviation); unit: years] | 34.7 (12.2) | 33.7 (12.0) | 35.3 (14.2) | 34.6 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 21 | 20 | 66
  Male | 38 | 38 | 39 | 115
Region of Enrollment [Number; unit: participants]
  United States | 37 | 34 | 34 | 105
  Canada | 26 | 25 | 25 | 76

OUTCOME MEASURES:

1. Primary Outcome: Rates of Remission (LSAS≤30) After 12 Weeks of Randomized Treatment During Phase II, Among Phase I Non-responders
Description: The Liebowitz Social Anxiety Scale (LSAS) is a 24-item scale assessing fear and avoidance in social and performance situations; it is widely used in studies of pharmacological treatment of Generalized Social Anxiety Disorder (GSAD). Scores on the LSAS range from 0 to 144, with higher scores indicating greater pathology.
Time Frame: Measured at Week 22 (Endpoint)
Population: The present analysis was conducted in the modified ITT population (n=181), with remission based on week 22 LSAS for study completers (n=154, and last Phase II LSAS for the 27 patients who terminated early.
Measure: Number; unit: participants
Arm/Group | Sertraline and Clonazepam | Venlafaxine | Sertraline and Placebo
Number analyzed (Participants) | 63 | 59 | 59
participants | 17 | 11 | 10

2. Secondary Outcome: Post-treatment Social Phobia Severity as Defined by Endpoint LSAS Scores
Description: The Liebowitz Social Anxiety Scale (LSAS) is a 24-item scale assessing fear and avoidance in social and performance situations; it is widely used in studies of pharmacological treatment of Generalized Social Anxiety Disorder (GSAD). We analyzed the overall change in LSAS (last Phase II LSAS minus Week 10 LSAS). Higher numbers reflect greater drops in social anxiety disorder severity. Scores on the LSAS range from 0 to 144, with higher scores indicating greater pathology.
Time Frame: Change from Week 10 to Week 22
Population: This analysis was conducted in Phase I non-responders, randomized to receive 12 weeks of continued sertraline plus the addition of clonazepam, switch to venlafaxine, or prolonged sertraline plus placebo.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sertraline and Clonazepam | Venlafaxine | Sertraline and Placebo
Number analyzed (Participants) | 63 | 59 | 59
units on a scale | 27 (24.4) | 18 (19) | 16 (23)

ADVERSE EVENTS:
Time Frame: Phase II, consisting of 12 weeks of randomized treatment.
Description: Patients were asked about the occurrence of adverse events during each visit. These will be recorded by the clinician on the Adverse Events form and rated as mild, moderate or severe.
Arm/Group | Sertraline and Clonazepam | Venlafaxine | Sertraline and Placebo
Serious Adverse Events (participants affected / at risk) | 3/63 | 0/59 | 0/59
Other Adverse Events (participants affected / at risk) | 51/63 | 51/59 | 55/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sertraline and Clonazepam (N=63) | Venlafaxine (N=59) | Sertraline and Placebo (N=59)
Shortness of Breath (General disorders) | 1 (1) | 0 (0) | 0 (0)
Panic Attack (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pacemaker inserted (General disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sertraline and Clonazepam (N=63) | Venlafaxine (N=59) | Sertraline and Placebo (N=59)
ASTHENIA (General disorders) | 11 (14) | 8 (10) | 15 (16)
HEADACHE (General disorders) | 12 (14) | 8 (11) | 15 (28)
ANOREXIA (General disorders) | 8 (9) | 11 (11) | 8 (9)
DRY MOUTH (General disorders) | 8 (8) | 12 (12) | 8 (8)
INSOMNIA (General disorders) | 8 (10) | 21 (27) | 25 (31)
LIBIDO DECREASED (General disorders) | 9 (9) | 6 (6) | 14 (15)
SOMNOLENCE (General disorders) | 20 (26) | 9 (11) | 14 (18)
ABNORMAL DREAMS (General disorders) | 6 (6) | 9 (9) | 11 (11)
ABNORMAL EJACULATION (General disorders) | 7 (8) | 6 (6) | 3 (3)
AMNESIA (General disorders) | 1 (1) | 3 (3) | 1 (1)
ANXIETY (General disorders) | 3 (3) | 1 (1) | 3 (3)
CONSTIPATION (General disorders) | 1 (1) | 6 (8) | 4 (5)
COUGH INCREASED (General disorders) | 2 (2) | 0 (0) | 3 (3)
DEPRESSION (General disorders) | 2 (2) | 4 (4) | 2 (2)
DIARRHEA (General disorders) | 7 (8) | 5 (5) | 11 (14)
DIZZINESS (General disorders) | 6 (6) | 7 (7) | 6 (6)
DYSPEPSIA (General disorders) | 3 (3) | 1 (1) | 5 (8)
INCREASED APPETITE (General disorders) | 2 (2) | 1 (1) | 4 (4)
INFECTION (General disorders) | 4 (5) | 5 (5) | 3 (3)
NAUSEA (General disorders) | 8 (8) | 7 (7) | 9 (11)
NERVOUSNESS (General disorders) | 4 (5) | 9 (11) | 10 (14)
PAIN (General disorders) | 2 (2) | 1 (1) | 5 (5)
PHARYNGITIS (General disorders) | 4 (4) | 3 (3) | 3 (4)
RASH (General disorders) | 1 (1) | 2 (2) | 3 (3)
SEXUAL FUNCTION ABNORMAL (General disorders) | 8 (8) | 6 (7) | 12 (14)
SWEATING (General disorders) | 1 (1) | 8 (8) | 10 (10)
THINKING ABNORMAL (General disorders) | 3 (3) | 2 (2) | 4 (4)
TOOTH DISORDER (General disorders) | 2 (2) | 5 (5) | 6 (7)
TREMOR (General disorders) | 6 (6) | 6 (6) | 2 (2)
TWITCHING (General disorders) | 1 (1) | 2 (2) | 4 (4)
URINARY FREQUENCY (General disorders) | 0 (0) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No